CLINICAL TRIAL: NCT03364582
Title: Dietary Patterns, Metabolomics and Colorectal Cancer Risk and Mortality in the Nurses' Health Study and Health Professionals Follow-Up Study
Brief Title: Dietary Patterns, Metabolomics and Colorectal Cancer Risk
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Fred Tabung, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-19280
Record Dates: First submitted 2017-11-27; First posted 2017-12-06 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer; Mortality
Keywords: Dietary patterns; Metabolomics; Mortaltiy; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples to analyze for inflammatory, insulin response biomarkers and metabololites
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men-observed dietary pattern: Health Professionals Follow-up Study: a prospective cohort of male health professionals
  Interventions: Other: Observed dietary pattern
- Women-observed dietary pattern: Nurses' Health Study: a prospective cohort of female registered nurses
  Interventions: Other: Observed dietary pattern

INTERVENTIONS:
Other: Observed dietary pattern — No intervention will be used. This is an observational study with dietary patterns as main exposure

SUMMARY:
Colorectal cancer (CRC) is the third most commonly diagnosed cancer in American men and women with ≥130,000 new cases each year. Several dietary patterns have been associated with CRC risk but underlying mechanisms are not fully understood. Researchers thus propose to integrate dietary patterns and metabolomics data to comprehensively investigate biological pathways linking dietary patterns and CRC risk.

DETAILED DESCRIPTION:
Several dietary patterns have been associated with colorectal cancer (CRC) risk but underlying mechanisms are not fully understood. Also, evidence is lacking on the consistency of dietary guidelines for overall health and CRC prevention given that it is not feasible to have an optimal diet for every disease. Furthermore, metabolomic profiling has not been widely assessed with respect to CRC risk. Metabolomics is uniquely suited to assess metabolic responses to dietary stimuli, given that it is situated downstream to all the other "omics". Building on prior work in hypothesis-driven dietary patterns and CRC prevention, the researchers seek to fill these knowledge gaps by proposing to: 1) use a standardized methodology to compare the best diet for overall health with the best diet for CRC prevention, and further determine if any associations of dietary patterns with CRC prevention are mediated by mechanisms involving inflammation and insulin; 2) determine metabolites that may mediate the association of dietary intake with CRC risk. The researchers will utilize two large prospective cohort studies, the Nurses' Health Study (NHS) and the Health Professionals Follow-up Study (HPFS), in which dietary and nondietary data have been collected every 2 to 4 years among 173,230 women and men over the last ≥30 years, with ≥3,400 CRC cases and ≥43,800 all-cause deaths. This integrated interrogation of dietary patterns and metabolomics data will inform the design of guidelines for healthful lifestyles that are optimized for CRC prevention.

ELIGIBILITY:
Inclusion Criteria:

-Adult health professionals

Exclusion Criteria:

* Any cancer except nonmelanoma skin cancer
* Did not complete a food frequency questionnaire during follow-up
* Had implausible values for total energy intake (<600 or >3500 kcal/d for women and <800 or >4,200 kcal/d for men) at study entry

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Nurses' Health Study (NHS) and the Health Professionals Follow-up Study (HPFS). The NHS recruited 121,701 registered female nurses aged 30 to 55 years at baseline in 1976, and the HPFS enrolled 51,529 male health professionals aged 40 to 75 years at baseline in 1986 in the United States. In both cohorts, questionnaires were sent at baseline and every two years thereafter to collect and update demographic, lifestyle, medical, and other health-related information. Since the inception of both cohorts, participants have completed self-administered questionnaires every 2 years, providing updated information on medical and lifestyle factors. Every 2 to 4 years, participants receive validated semi-quantitative food frequency questionnaires (FFQ) for dietary assessments.
Sampling Method: Non-Probability Sample
Enrollment: 173230 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Colorectal cancer risk | 1986 to 2012 (men), 1984 to 2012 (women)
  Incident colorectal cancer

SECONDARY OUTCOMES:
incident total cardiovascular disease, total cancer, chronic respiratory diseases | 1986 to 2012 (men), 1984 to 2012 (women)
  The incidence of these major chronic diseases will be examined as surrogate for overall health
Mortality | 1986 to 2012 (men), 1984 to 2012 (women)
  Incident death of any cause (as surrogate for overall health)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Tabung, PhD, MSHP, Principal Investigator — Ohio State Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee DH, Jin Q, Shi N, Wang F, Bever AM, Li J, Liang L, Hu FB, Song M, Zeleznik OA, Zhang X, Joshi A, Wu K, Jeon JY, Meyerhardt JA, Chan AT, Eliassen AH, Clish CB, Clinton SK, Giovannucci EL, Tabung FK. Dietary Inflammatory and Insulinemic Potentials, Plasma Metabolome and Risk of Colorectal Cancer. Metabolites. 2023 Jun 12;13(6):744. doi: 10.3390/metabo13060744. PMID 37367904
- [Result] Lee DH, Jin Q, Shi N, Wang F, Bever AM, Liang L, Hu FB, Song M, Zeleznik OA, Zhang X, Joshi A, Wu K, Jeon JY, Meyerhardt JA, Chan AT, Eliassen AH, Clish C, Clinton SK, Giovannucci EL, Li J, Tabung FK. The metabolic potential of inflammatory and insulinaemic dietary patterns and risk of type 2 diabetes. Diabetologia. 2024 Jan;67(1):88-101. doi: 10.1007/s00125-023-06021-3. Epub 2023 Oct 11. PMID 37816982
- [Derived] Petimar J, Smith-Warner SA, Fung TT, Rosner B, Chan AT, Hu FB, Giovannucci EL, Tabung FK. Recommendation-based dietary indexes and risk of colorectal cancer in the Nurses' Health Study and Health Professionals Follow-up Study. Am J Clin Nutr. 2018 Nov 1;108(5):1092-1103. doi: 10.1093/ajcn/nqy171. PMID 30289433
- [Derived] Tabung FK, Wang W, Fung TT, Smith-Warner SA, Keum N, Wu K, Fuchs CS, Hu FB, Giovannucci EL. Association of dietary insulinemic potential and colorectal cancer risk in men and women. Am J Clin Nutr. 2018 Aug 1;108(2):363-370. doi: 10.1093/ajcn/nqy093. PMID 29901698
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03364582/Prot_SAP_000.pdf